CLINICAL TRIAL: NCT00664872
Title: Effect of Proactive Psychosocial Treatment by the Case Manager in Patients After a Suicide Attempt: a Randomised Controlled Trial
Brief Title: Effect of Psychosocial Treatment by the Case Manager in Patients After a Suicide Attempt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shen-Ing,Liu (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Shen-Ing,Liu, Attending Physician, Mackay Memorial Hospital
Organization: Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC96-2314-B195-011
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Suicide, Attempted
Keywords: case manager; suicide; attempt; effectiveness
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- case management (Experimental)
  Interventions: Other: proactive psychosocial intervention by care managers; Behavioral: case management

INTERVENTIONS:
Other: proactive psychosocial intervention by care managers — A case manager will be assigned to each of the participants in the intervention group. All case managers are psychologists. After discharge from the emergency department, the participants receive six sessions of proactive psychosocial intervention by their case manager over four months. Duration of each session is approximately 30 minutes. The intervention consists of telephone or face-to-face contacts with the case manager at scheduled intervals or when clinically necessary. If a patient declines medication therapy from the psychiatrist, case manager will provide psychotherapy using the model of cognitive-behavioural approach and problem-solving therapy. Case managers will receive backup and supervision by psychiatrist investigators and monthly supervision of therapy. Case managers will regularly monitor suicide risk, clinical status and provide follow-up.
Behavioral: case management

SUMMARY:
The purpose of this study is to determine the case manager are effective in the treatment of suicide attempters.

DETAILED DESCRIPTION:
Compared with usual care, interventional group will (1) improve treatment attendance, (2) have less repeated suicide attempts in adults after a suicide attempts, and (3)have better patients' satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

Participants recruit adults who:

1. Discharge from an emergency department of a teaching hospital after attempt suicide
2. Aged above 18 years old
3. Agree to provide written inform consent.

Exclusion Criteria:

1. Patients were too ill to be interviewed
2. Patients have immediate and severe suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
treatment adherence, defined as outpatient mental health clinic attendance | 6-month, and 12-month

SECONDARY OUTCOMES:
During follow-up periods (6-month, and 12-month), interventional group will have (1) less repeated suicide attempts (behavior) (2) less suicidal ideation, (3) lower depression score, (4) better patients' satisfaction with care | 6-month, and 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Shen-Ing Liu, MD.PHD, Principal Investigator — Department of Psychiatry, Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617